CLINICAL TRIAL: NCT01693445
Title: Dose Finding Study of S-1, Oxaliplatin, and Irinotecan Combination Chemotherapy for Patients With Inoperable Advanced or Metastatic Gastrointestinal Cancers
Brief Title: S-1, Oxaliplatin, and Irinotecan for Advanced Gastrointestinal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hallym University Medical Center (Other)
Collaborators: Jeil Pharmaceutical Co., Ltd. (Industry); HK inno.N Corporation (Industry); Pfizer (Industry); Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMC-HO-GI-1203
Record Dates: First submitted 2012-09-20; First posted 2012-09-26 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2012-09

CONDITIONS: Gastrointestinal Neoplasms
Keywords: Gastrointestinal neoplasms; Oxaliplatin; Irinotecan; S-1
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — Oxaliplatin; Irinotecan; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OIS (Oxaliplatin, Irinotecan, S-1) (Experimental): Dose level 1 treatment will be delivered as a 2-week cycle as bellows;
  1. Oxaliplatin 85 mg/m²IV on day 1
  2. Irinotecan 120 mg/m² IV on day 1
  3. S-1 60 mg/m2/day PO on day 1-7 Dose escalation will be continued until more than one-third of the patients in a given cohort show dose limiting toxicities (DLT) during treatment cycle 1. If at least 2 patients are observed to have DLT, this dose level is defined as the maximum tolerated dose (MTD). If exactly 1 of the 3 patients treated show DLT, 3 additional patients are treated at the current dose level.
  Interventions: Drug: OIS (Oxaliplatin, Irinotecan, S-1)

INTERVENTIONS:
Drug: OIS (Oxaliplatin, Irinotecan, S-1) — Dose level 1 treatment will be delivered as a 2-week cycle as bellows;
  1. Oxaliplatin 85 mg/m²IV on day 1
  2. Irinotecan 120 mg/m² IV on day 1
  3. S-1 60 mg/m2/day PO on day 1-7
  Dose escalation will be continued until more than one-third of the patients in a given cohort show dose limiting toxicities (DLT) during treatment cycle 1. If at least 2 patients are observed to have DLT, this dose level is defined as the maximum tolerated dose (MTD). If exactly 1 of the 3 patients treated show DLT, 3 additional patients are treated at the current dose level.
  Other Names: Kabioxaliplatin; Campto; TS-1

SUMMARY:
This study will attempt to determine the feasibility of combination of Oxaliplatin, Irinotecan, and S-1, the maximum tolerated dose and the recommended doses of the agents used, and to preliminarily evaluate the antitumor activity in untreated patients with advanced gastrointestinal cancer.

DETAILED DESCRIPTION:
Oxaliplatin or irinotecan has shown a considerable anti-tumor activity, when used in combination with 5-fluorouracil (5-FU) in patients with gastrointestinal (GI) cancer. Oxaliplatin, irinotecan, and 5-FU have different mechanisms of actions and do not share the toxicity profiles. Since they have a synergistic effect, many clinical trials have been conducted recently to evaluate the efficacy of triplet combination consisting of oxaliplatin, irinotecan, and 5-FU, and demonstrated that the triple combination regimen was effective and resulted in survival benefits with favorable toxicity profiles.

S-1 and capecitabine are novel oral fluoropyrimidines and different phase III trials have shown that these oral agents are at least as active and effective as 5-FU with a superior safety profile.

Biweekly triple combination of S-1 with oxaliplatin and irinotecan (OIS) is an interesting alternative to increase convenience and to simply the treatment delivery.

In the present study, we attempt to determine the feasibility of OIS combination, the maximum tolerated dose and the recommended doses of the agents used, and to preliminarily evaluate the antitumor activity in untreated patients with advanced gastrointestinal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven recurrent or metastatic adenocarcinoma of the gastrointestinal tract
* Minimum age of 18 years
* ECOG Performance status 0-2
* Life expectancy >3 months
* Presence of measurable or evaluable disease by RECIST
* Prior adjuvant chemotherapy without S-1, oxaliplatin and irinotecan is allowed if more than 4 weeks elapsed since completion of chemotherapy.
* More than 4 weeks since completion of prior radiotherapy (measurable or evaluable lesions should be outside the radiation field)
* Adequate organ functions
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study in keeping with the policy of the hospital

Exclusion Criteria:

* Patients treated previously with S-1, oxaliplatin, or irinotecan as adjuvant chemotherapy.
* Patients with CNS metastases or carcinomatous leptomeningitis or neurologic disease.
* Patients with active infection, severe heart disease, uncontrollable hypertension or diabetes mellitus, myocardial infarction during the preceding 6 months, pregnancy, or breast feeding
* Any previous or concurrent malignancy other than non-melanoma skin cancer or in situ cancer of uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2012-06; Primary Completion 2014-02 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
maximum tolerated dose | 6 months

SECONDARY OUTCOMES:
toxicity profiles | 6 months
overall response rate | 6 months
progression free survival | 6 months
overall survival | 6 months
disease control rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dae Young Zang, MD, PhD, Principal Investigator — Hallym University Medical Center
Locations (1):
- Hallym University Medical Center, Anyang, South Korea

IPD SHARING:
Plan to Share IPD: Undecided